CLINICAL TRIAL: NCT07337499
Title: Comparison of the Maglumi X3 SNIBE Method With Other Analytical Methods in Laboratory Medicine
Brief Title: Comparison of Maglumi X3 SNIBE With Other Analytical Methods in Laboratory Medicine for 25-(OH)D Quantification
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Snibe(L4174)
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-03

CONDITIONS: Quantification of 25-(OH)D in Physiological Condition
Keywords: 25-(OH)D; vitamin D; analytical methods; immunoassay
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 200 subjects: healthy volunteers and patients scheduled for orthopedic and cardiothoracic surgery: Two hundred subjects will include healthy volunteer individuals, employees of the Galeazzi-Sant'Ambrogio Hospital, and patients at the time of pre-admission or admission who are scheduled for major orthopedic surgery involving hip or knee prostheses, or for cardiothoracic surgery, as these represent the largest cohorts within our institution. All subjects will be older than 18y, without cancer, obesity, not pregnant, and able to understand or make decisions.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — No intervention, besides blood sampling for 25-(OH) vitamin D quantification, is required since this study intends to assess the agreement among the results obtained using the Maglumi X3 SNIBE method and other analytical methods for the measurement of 25-(OH) vitamin D.

SUMMARY:
The aim of this study is to assess the agreement among the results obtained using the Maglumi X3 SNIBE method and other analytical methods for the measurement of 25-(OH) vitamin D. The comparison between analytical methods is essential for evaluating the analytical performance of different measurement techniques. Assessing the level of comparability between measurements of the same analyte obtained using different methods is fundamental for the harmonization and quality of procedures used in laboratory medicine, ensuring a correct clinical interpretation of results.

DETAILED DESCRIPTION:
The analytical methods most commonly used in clinical laboratories and for which harmonization/standardization of procedures is required are immunoassays, which enable the quantification of an analyte.

Currently, the reference method for immunoassays is liquid chromatography tandem mass spectrometry (LC-MS/MS). LC-MS/MS is increasingly used in clinical laboratories. Its high specificity, sensitivity, and multi-analyte capability make it an ideal alternative to immunoassays or conventional high-performance liquid chromatography (HPLC). LC-MS/MS also provides greater flexibility than immunoassays, as LC-MS/MS assays are typically developed in-house. In addition, a single LC-MS/MS run can generate a large amount of quantitative or qualitative data.

All of these methods are essential in clinical diagnostics because they allow the detection and quantification of a wide range of biomarkers, including hormones, proteins, and antibodies across numerous areas of medicine. Despite their widespread use and importance, variability between different methods, within the same laboratory or across laboratories, represents a significant challenge, with considerable impact on results, clinical decisions, and ultimately on patient care. This variability may depend on various factors, including the quality and source of reagents, the quality of calibrators critical for analyte quantification, detection methods, and testing protocols.

Every clinical laboratory is therefore required to assess the agreement of results whenever new instruments or analytical procedures are introduced, compared with a method already in use. Method comparison is indeed one of the principals of the International Standard (ISO 15189:2012) for the accreditation of medical laboratories and of the IVD Directive 98/79 EC, which defines the requirements for in vitro diagnostic devices (IVDs) at the European level.

The comparison of two methods requires defining a maximum acceptable difference between the concentrations of an analyte obtained using the analytical techniques of interest; therefore, two methods may be considered comparable if the differences between the results are below a predefined acceptable limit: the maximum acceptable error. The definition of the maximum acceptable error is based on analytical quality specifications established according to five hierarchical models defined at the 1999 Stockholm Conference:

* a model based on the evaluation of the effect of analytical performance on clinical outcomes under specific clinical conditions;
* a model based on the evaluation of the effect of analytical performance on clinical decisions;
* a model based on the biological variability of the analyte;
* a model based on published expert recommendations;
* a model based on the current state of the art (of instruments and/or methods), derived for example from EQA programs.

Therefore, the study will be structured into several phases, beginning with the collection of information on the analytical characteristics and performance of the instruments being compared, verifying method repeatability. For each analyte, the maximum acceptable error will be defined a priori, based on analytical quality specifications, such as analytical imprecision and inaccuracy.

Statistical tests will be performed to assess the error between the analyte measurements obtained using the different methods and, if comparability is not achieved, additional evaluations will be carried out to rule out methodological errors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer subjects:

Subjects who sign the informed consent to participate in the study Age ≥ 18 years Employees, in various roles, of the IRCCS Galeazzi-Sant'Ambrogio Hospital

-Patients:

Subjects who sign the informed consent to participate in the study Age ≥ 18 years Patients referred for major orthopedic surgery: hip and knee replacement (bicompartmental and unicompartmental) Patients referred for cardiothoracic surgery

Exclusion Criteria:

* Neoplastic diseases (until remission)
* Grade I, II, and III obesity
* Age < 18 years
* Women who are pregnant or breastfeeding, based on self-declaration
* Individuals unable to understand and make decisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred subjects will be recruited, including healthy individuals who are employees of the Galeazzi-Sant'Ambrogio Hospital, as well as patients at the time of pre-admission or admission who are referred for major orthopedic surgery (hip and knee replacement) or for cardiothoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of 25-(OH) vitamin D quantification with LC-MS/MS and Maglumi X3 SNIBE | The study requires a single time point
  The primary outcome of this study is to evaluate the agreement between the results obtained for the measurement of 25-(OH) vitamin D using the Maglumi X3 SNIBE method and other analytical methods . Serum level of 25-(OH) vitamin D will be measured in 200 subjects enrolled in Ospedale Galeazzi-Sant'Ambrogio and than analyzed using appropriate statistic test to define the maximum acceptable error among the measurements.

SECONDARY OUTCOMES:
Comparison of 25-(OH) vitamin D quantification with Maglumi X3 SNIBE and other immunoassay based analytival methods | The study requires a single time point
  The secondary outcomes of this study are to evaluate the agreement among the results obtained for the measurement of 25-(OH) vitamin D using the Maglumi X3 SNIBE method and other analytical methods . Serum level of 25-(OH) vitamin D will be measured in 200 subjects enrolled in Ospedale Galeazzi-Sant'Ambrogio and than analyzed using appropriate statistic test to define the maximum acceptable error among the measurements obtained using the diffente methods

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Lombardi, PhD, Principal Investigator — IRCCS Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- Laboratory of Experimental Biochemistry and Advanced Diagnostic, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
The data generated in this study may be made available upon reasonable request after the primary results have been published.

REFERENCES:
- [Background] Fraser CG. The 1999 Stockholm Consensus Conference on quality specifications in laboratory medicine. Clin Chem Lab Med. 2015 May;53(6):837-40. doi: 10.1515/cclm-2014-0914. PMID 25720125
- [Background] Leung KS, Fong BM. LC-MS/MS in the routine clinical laboratory: has its time come? Anal Bioanal Chem. 2014 Apr;406(9-10):2289-301. doi: 10.1007/s00216-013-7542-5. Epub 2013 Dec 15. PMID 24337187
- [Background] Terzapulo X, Kassenova A, Bukasov R. Immunoassays: Analytical and Clinical Performance, Challenges, and Perspectives of SERS Detection in Comparison with Fluorescent Spectroscopic Detection. Int J Mol Sci. 2024 Feb 8;25(4):2080. doi: 10.3390/ijms25042080. PMID 38396756
- [Background] Plebani M. Harmonization in laboratory medicine: Requests, samples, measurements and reports. Crit Rev Clin Lab Sci. 2016;53(3):184-96. doi: 10.3109/10408363.2015.1116851. Epub 2015 Dec 15. PMID 26667798
- [Background] Zaninotto M, Graziani MS, Plebani M. The harmonization issue in laboratory medicine: the commitment of CCLM. Clin Chem Lab Med. 2022 Nov 16;61(5):721-731. doi: 10.1515/cclm-2022-1111. Print 2023 Apr 25. PMID 36383396